## Forespørsel om å delta i studien av molekylærbiologiske forandringer i svulstvev som kan forutsi behandlingseffekt

Som du er blitt informert om er brystkreftsvulsten din av en slik type at vi anbefaler behandling med cellegift før operasjon. Vi har praktisert slik behandling ved vår avdeling i 15 år og tilsvarende behandlingsprinsipper brukes ved alle norske universitetssykehus og de aller fleste sykehus i den vestlige verden det er naturlig for oss å sammenligne oss med.

Utgangspunktet er at ved svulster som din viser all klinisk erfaring at det er nødvendig å gi cellegift i tillegg da dette vil kunne forebygge senere tilbakefall. Tradisjonelt har denne vært gitt etter operasjonen. Fordelen med å gi den før operasjonen er imidlertid at man legger forholdene bedre til rette for kirurgi. Samtidig får vi da en mulighet til direkte å måle effekten av cellegiften, hvilket betyr at dersom den ikke virker slik vi ønsker har vi muligheten til å skifte til et annet medikament.

I din situasjon ønsker vi å gi deg behandling med to ulike typer cellegift, hver gitt over en 8 ukers periode. Å gi hvert enkelt medikament alene byr på fordeler fremfor å gi dem kombinert. På denne måten kan vi gi de riktige doser av hvert av medikamentene uten at dette gir uakseptable bivirkninger. På den andre siden ønsker vi å gi medikamentet noe hyppigere (hver 14. dag) enn det som ellers er vanlig nemlig hver 3. uke. Dette er basert på en stor studie fra USA der man ga et tilsvarende regime til pasienter etter operasjon. I dette tilfellet viste det seg at det i større grad forebygde tilbakefall. Tatt i betraktning av at svulsten din er relativ stor ønsker vi å tilby deg behandling med et slikt noe mer "intensivt" regime da vi mener dette er den beste behandlingsform vi per i dag kjenner til.

Forskningsdelen i denne studien ligger i at vi ønsker å undersøke molekylære forandringer i svulstvevet som kan ha sammenheng med behandlingseffekt. Det er velkjent at samme behandlingsregime har ulik effekt på svulstene hos forskjellige pasienter. Vi vet per i dag ikke sikkert grunnen til dette. Kan vi finne mer ut av disse mekanismene åpner det for muligheten til å "skreddersy" behandling til hver enkelt pasient i fremtiden, idet vi da på grunnlag av en prøve kan forutsi hvilket medikament den enkelte vil ha størst nytte av. Forhåpentligvis vil slike resultater på sikt kunne åpne muligheten for at vi også skal kunne helbrede svulster vi ikke kan kurere i dag.

Rent praktisk vil deltakelse i denne studien innebære for deg at vi vil ta ut noe ekstra vev før behandling for å ha til vitenskapelige studier. Vanlig klinisk rutine er at vi med en grov nål vil ta ut et par mindre vevsbiter før behandlingsstart for å bekrefte diagnose. Dersom du er villig til å delta i studien vil vi i stedet for sette lokalbedøvelse og skjære ut en liten bit av svulstvevet som både gir oss mulighet til endelig bekreftelse av diagnose samt kunne brukes til å gjennomføre de spesialundersøkelser vi ønsker i vårt forskningsprosjekt. I tillegg vil vi, dagen etter første cellegiftbehandling ved begge regimene og når du etter 8 ukers behandling skifter fra det ene medikamentet til det andre, ta en ny vevsprøve da med en grov nål. Til slutt vil vi når du behandles med operasjon ta ut noe av vevet og bruke til våre forskningsstudier.

I våre undersøkelser ønsker vi å kartlegge hvilke forandringer som foreligger i selve svulstvevet. Slike forandringer opptrer i alle kreftsvulster og har som regel ikke noe med nedarvet disposisjon å gjøre. Når vi imidlertid finner en genforandring i svulstvevet ønsker vi å være sikker på at den ikke samtidig finnes i normal-vevet i kroppen. Av den grunn tar vi også en blodprøve fra deg for å undersøke om de samme genforandringer er tilstede i de hvite blodlegemer. Det er således en teoretisk risiko for at man kan komme til å finne en nedarvet gen-disposisjon hos enkelte individer som deltar i en studie som denne, selv om den risikoen er liten. Dersom vi skulle finne en slik forandring vil vi normalt ikke gå ut med informasjon til deg om den. Du står imidlertid til enhver tid fritt å spørre om vi har foretatt slike genanalyser og i tilfelle hva som har vært resultat av disse.

Det understrekes at deltakelse i studien er frivillig og du har anledning til når som helst å trekke deg dersom du måtte ønske dette uten at du trenger å gi noen begrunnelse for det. I dette ligger at dersom du har avgitt vev kan du kreve at alle opoplysninger blir anonymisert så ingen kan identifisere at vevet kommer fra deg.

Vi har planlagt å utføre laboratorie-arbeidet i vårt eget forskningslaboratorium, eventuelt i samarbeide med andre forsknings-grupper i Norge. Med tanke på enkelte spesial-analyser, kan det bli aktuelt å samarbeide med utenlandske laboratorier med spesial-kompetanse; i så fall vil vi sende litt materiale dit. Dersom dette skulle bli aktuelt, vil materialet bli merket på en slik måte at det ikke er mulig for noen av forskerne i utlandet å finne fram til din identitet. Vi er imidlertid lov-pålagt å informere deg om at slik utførsel muligens er aktuelt, i og med at du har anledning til å nekte dette.

Studien er godkjent av Den Regionale Komite for Madisinsk Forskningsetikk, Sosial og Helsedirektoratet (Lov om Opprettelse av Biobank) samt datatilsynet via Norsk samfunnsvitenskapelig Datatjeneste.

Prosjektet gjennomføres i regi av Helse-Bergen ved Kreftavdelingen, haukeland Sykehus. Ansvarlig prosjektleder er Professor / Overlege Per Eystein Lønning ved Kreftavdelingen. Prosjektet varer fram til 1/9-2020, men det er mulig at man fortsatt vil analysere data etter dette.

Dersom du ikke skulle ønske å delta i denne studien vil du få vanlig standard behandling som også innebærer at vi tilbyr cellegiftbehandling før operasjon med et noe annet regime enn det som er foreslått her.

Per Eystein Lønning, Professor Dr. Med, Kreftavdelingen, Haukeland Sykehus

| Undertegnede har lest ovenstående informasjon. |
|------------------------------------------------|
| Jeg sier meg villig til å delta i studien: |
| Dato |